CLINICAL TRIAL: NCT04569539
Title: The Effect of a Head Elevated Positioning Device on Position, Height and Depth of the Cricothyroid Membrane in Morbidly Obese Pregnant Women in the Third Trimester.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-02
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Airway Complication of Anesthesia
Keywords: cricothyroid membrane; pregnancy; obesity; ultrasound
MeSH Terms: conditions — Obesity | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Experimental): Ultrasound measurements of the cricothyroid membrane
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound scan of the cricothyroid membrane

SUMMARY:
The cricothyroid membrane (CTM) is situated in the anterior neck and may be readily palpated in most people. In the event of difficulties securing the airway during a general anesthetic the CTM can facilitate emergency access to the upper airway to allow rescue oxygenation and ventilation. Caesarean sections are today carried out using either a spinal or epidural anaesthesia and for good reason. Due to physiological effects of pregnancy a patient's airway is known to be more challenging when pregnant than outside of pregnancy. The pregnant airway can even change over the course of labor. Airway ultrasound has become increasingly popular and allows accurate identification of airway structures including the cricothyroid membrane. It has already shown to be more accurate than palpation alone in identifying the cricothyroid membrane in obese pregnant women. The incidence of obesity in pregnancy continues to increase. Although regional anesthesia is preferred when these women require Caesarean section this is not always possible or successful. Use of a device to optimise patient position for airway management is the standard of practice for obese pregnant patients. These devices are known as head elevating laryngoscopy position pillows, the TROOP elevation pillow ® is one such device. However, the investigators do not know if and how positioning the obese pregnant patient on a TROOP elevation pillow ® affects position, depth and height of the cricothyroid membrane. The investigators want to know if the TROOP elevation pillow ® will hinder or facilitate the performance of a surgical airway in the event of failed airway management in the pregnant obese patient.

The investigators hypothesize that in pregnant obese patients in the third trimester use of the TROOP elevation pillow ® will change the position, height and depth of the CTM compared to the neutral position. Based on previous evidence the investigators believe the position of the membrane will move superiorly in relation to the sternal notch, will increase in height and the depth from the skin to the membrane will be reduced. The investigators also hypothesize that CTM identification and marking prior to final patient positioning may be misleading.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients in third trimester (>28/40 weeks)
* Morbid Obesity (BMI≥40kg/m2)
* Ability to understand the rationale of the study assessments and to provide signed consent - Ability to safely and comfortably take part in the study protocol

Exclusion Criteria:

* Non pregnant patients
* Pregnant patients less than 28 weeks pregnant
* Not Morbidly Obese (BMI≥40kg/m2)
* Cervical spine pathology causing restricted neck movement or neurological compromise - Previous neck surgery or irradiation
* Upper limb neurology
* Patient refusal

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
The change in the CTM midpoint between neutral positioning and the head elevated position. | 10 min
  The head will be elevated using the TROOP elevating pillow ®.

SECONDARY OUTCOMES:
The change in depth of the CTM between neutral positioning and the head elevated. | 10 min
  The head will be elevated using the TROOP elevating pillow ®.
The change in height of the CTM between neutral positioning and the head elevated. | 10 min
  The head will be elevated using the TROOP elevating pillow ®.
The change in distance from the sternal notch to the CTM mid-point between neutral positioning and the head elevated. | 10 min
  The head will be elevated using the TROOP elevating pillow ®.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No